CLINICAL TRIAL: NCT06809699
Title: A Prospective Single-arm Trial on Human Leukocyte Antigen (HLA) Mismatched Related Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Human Leukocyte Antigen (HLA) Mismatched Related Allogeneic Hematopoietic Stem Cell Transplantation
Acronym: HIGHT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: He Huang (Other)
Responsible Party: Sponsor-Investigator, He Huang, Professor, Director of the Bone Marrow Transplantation Center, The First Affiliated Hospital, Zhejiang University School of Medicine, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMR-001
Record Dates: First submitted 2024-10-04; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-10

CONDITIONS: Hematologic Diseases
Keywords: Hematopoietic cell transplantation; HLA mismatch related; Hematologic diseases
MeSH Terms: conditions — Hematologic Diseases | interventions — Busulfan; Cyclophosphamide; fludarabine; fludarabine phosphate; Semustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HLA-mismatch related (Experimental): The myeloablative conditioning is used when the patient is below 50 and with an HCT-CI<2. The reduced intensity conditioning is used when the patient is over 50 or with an HCT-CI≥2.
  Interventions: Drug: Busulfan (Busulfex); Drug: Cyclophosphamide (CTX); Drug: Fludarabine (Fludara); Drug: Semustine (MeCCNU)

INTERVENTIONS:
Drug: Busulfan (Busulfex) — For myeloablative conditioning: Busulfan (Bu，3.2 mg/kg/d IV -8d ~-6d) For reduced intensity conditioning: (Bu，3.2 mg/kg/d IV -7d~-5d)
Drug: Cyclophosphamide (CTX) — Cyclophosphamide is only used in myeloablative conditioning (Cy，1.8g/m2, -5d, -4d)
Drug: Fludarabine (Fludara) — For myeloablative conditioning: Fludarabine (Flu，30 mg/m2/d IV -6d ~ -2d) For reduced intensity conditioning: Fludarabine（Flu，30mg/m2 /d IV -10d~-5d）
Drug: Semustine (MeCCNU) — For both myeloablative and reduced intensity conditioning: Semustine (MECCNU，250 mg/m2 orally-3d).

SUMMARY:
This study is a single center, prospective, single arm exploratory clinical trial that includes patients with hematological malignancies who are indicated for allogeneic hematopoietic stem cell transplantation (allo HSCT) but lack suitable donors. This project plans to use human leukocyte antigen (HLA) mismatched donors. Ultimately, a HLA mismatched allo HSCT transplantation plan will be established to improve the disease prognosis of these patients and truly enter the era of "everyone has a donor".

DETAILED DESCRIPTION:
This study is a single center, prospective, single arm exploratory clinical trial that includes patients with hematological malignancies who are indicated for allogeneic hematopoietic stem cell transplantation (allo HSCT) but lack suitable donors. This project plans to use human leukocyte antigen (HLA) mismatched donors. Ultimately, a HLA mismatched allo HSCT transplantation plan will be established to improve the disease prognosis of these patients and truly enter the era of "everyone has a donor".

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-60 years old) with hematological malignancies and indications for hematopoietic stem cell transplantation with no available related human leukocyte antigen (HLA) identical sibling donors;
* No available donor with HLA high-resolution typing ≥ 9/10 or those who have difficulty finding donors due to urgent medical conditions;
* No suitable HLA matching haploidentical donor available;
* There is a suitable donor with mismatched HLA typing;
* The subjects or their legal representatives shall sign an informed consent form before the start of the clinical study.

Exclusion Criteria:

* Patients with severe liver and kidney function (alanine aminotransferase>2.5 times the upper limit of normal, blood creatinine>1.5 times the upper limit of normal) and cardiopulmonary dysfunction (New York Heart Association (NYHA) III/IV heart function, ejection fraction<50%, severe obstructive or restrictive ventilation dysfunction);
* Merge active infections;
* Eastern Cooperative Oncology Group (ECOG) score ≥ 2 points;
* Secondary tumors with merged activity;
* Severe central nervous system or mental illness leading to the inability to autonomously choose to enter or exit clinical trials;
* Combine other allo HSCT contraindications.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1-year
  Overall survival after allogeneic cell transplantation refers to the length of time a patient remains alive from the date of transplantation, regardless of disease status or complications.

SECONDARY OUTCOMES:
Neutrophil engraftment rate | 28 days
  The neutrophil engraftment rate is assessed, and neutrophil engraftment is defined as achievement of an absolute neutrophil count (ANC) of ≥ 0.5 × 10⁹/L for three consecutive days
Platelet engraftment rate | 28 days
  Platelet engraftment rate is assessed, and platelet engraftment is defined as achievement of a platelet count of ≥ 20 × 10⁹/L (or ≥ 50 × 10⁹/L in some definitions) without transfusion support for at least seven consecutive days.
Relapse | 1-year
  Cumulative incidence of relapse
Cumulative incidence of relapse | 1-year
  Progression-free survival after allogeneic cell transplantation refers to the length of time during which a patient remains alive without any signs of disease relapse or progression.
Progression free survival | 1-year
  Progression-free survival after allogeneic cell transplantation refers to the length of time during which a patient remains alive without any signs of disease relapse or progression.
GRFS | 1-year
  GRFS (Graft-versus-host disease-free, relapse-free survival) after allogeneic cell transplantation is the length of time a patient remains alive without experiencing significant graft-versus-host disease, disease relapse, or death.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, China, China

IPD SHARING:
Plan to Share IPD: No